CLINICAL TRIAL: NCT02618304
Title: Changes of Tear-film Lipid Layer Thickness and Ocular Aberration After Treatment of Meibomian Gland Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-2015-0012
Record Dates: First submitted 2015-11-18; First posted 2015-12-01 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Meibomian Gland Dysfunction
Keywords: Meibomian gland dysfunction; Lipiview; Tear Lipid Layer
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- moderate to severe meibomian gland dysfunction (Experimental)
  Interventions: Drug: Treatment of Meibomian gland dysfunction

INTERVENTIONS:
Drug: Treatment of Meibomian gland dysfunction — artificial tears, 3% Diquafosol Tetrasodium eye drops, steroid eye drops, squeezing of meibomian glands, cleansing of eyelids.

SUMMARY:
In this study, investigator aim to evaluate the changes of tear-film lipid layer thickness and ocular aberration after treatment of meibomian gland dysfunction. In case of stage 3 or 4 meibomian gland dysfunction, participants will be treated using conventional treatment modalities. Before treatment and after 1 and 2 months of treatment, a variety of ophthalmic examination, tear-film lipid layer thickness, and ocular aberration are going to measured and compared.

ELIGIBILITY:
Inclusion Criteria:

1. age over 19 years old, with moderate to severe Meibomian gland dysfunction.

Exclusion Criteria:

1. patients with history of previous ocular or intraocular surgery
2. ocular infection, non dry eye ocular inflammation, ocular allergy, autoimmune disease
3. history of intolerance or hypersensitivity to any component of the study medications
4. wearing contact lenses during the study period, presence of current punctal occlusion
5. pregnancy, lactating women, and children

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2016-02-19 (Actual); Study Completion 2016-02-19 (Actual)

PRIMARY OUTCOMES:
Changes of tear-film lipid layer thickness after treatment of meibomian gland dysfunction | 1 and 2 months after treatment of meibomian gland dysfunction
Changes of ocular aberration after treatment of meibomian gland dysfunction | 1 and 2 months after treatment of meibomian gland dysfunction
  ocular parameters measured by Ray-tracing wavefront aberrometers (i-Trace, Tracey technologies , Texas ,USA)

SECONDARY OUTCOMES:
Corneal erosion grade(oxford score) | 1 and 2 months after treatment of meibomian gland dysfunction
OSDI(ocular surface disease index) | 1 and 2 months after treatment of meibomian gland dysfunction
Meibomian gland abnormality | 1 and 2 months after treatment of meibomian gland dysfunction
  measured by physiological parameter (score 0,1,2,3,4)
Meibomian quality | 1 and 2 months after treatment of meibomian gland dysfunction
  measured by physiological parameter (score 0,1,2,3,4)
BUT(tear break-up time) | 1 and 2 months after treatment of meibomian gland dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Yonsei Univeristy College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Asbell PA, Stapleton FJ, Wickstrom K, Akpek EK, Aragona P, Dana R, Lemp MA, Nichols KK. The international workshop on meibomian gland dysfunction: report of the clinical trials subcommittee. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):2065-85. doi: 10.1167/iovs.10-6997h. Print 2011 Mar. No abstract available. PMID 21450920
- [Background] Geerling G, Tauber J, Baudouin C, Goto E, Matsumoto Y, O'Brien T, Rolando M, Tsubota K, Nichols KK. The international workshop on meibomian gland dysfunction: report of the subcommittee on management and treatment of meibomian gland dysfunction. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):2050-64. doi: 10.1167/iovs.10-6997g. No abstract available. PMID 21450919
- [Background] Tomlinson A, Bron AJ, Korb DR, Amano S, Paugh JR, Pearce EI, Yee R, Yokoi N, Arita R, Dogru M. The international workshop on meibomian gland dysfunction: report of the diagnosis subcommittee. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):2006-49. doi: 10.1167/iovs.10-6997f. Print 2011 Mar. No abstract available. PMID 21450918
- [Background] McCulley JP, Shine WE. The lipid layer of tears: dependent on meibomian gland function. Exp Eye Res. 2004 Mar;78(3):361-5. doi: 10.1016/s0014-4835(03)00203-3. PMID 15106913